CLINICAL TRIAL: NCT00383370
Title: A Trial to Assess the Safety and Tolerability of Repeated Doses of Intravitreal Administration of Two VEGF Trap Formulations in Subjects With Neovascular Age Related Macular Degeneration
Brief Title: Safety and Tolerability of Intravitreal VEGF Trap Formulations in Subjects With Neovacular AMD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Avner Ingerman, MD, Regeneron Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VGFT-OD-0603
Record Dates: First submitted 2006-10-02; First posted 2006-10-03 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-04

CONDITIONS: Neovascular Age Related Macular Degeneration
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ITV-1 (Experimental): VEGF Trap formulation 1
  Interventions: Drug: VEGF Trap
- ITV-2 (Experimental): VEGF Trap formulation 2
  Interventions: Drug: VEGF Trap
- ITV-2 OL (Experimental): VEGF Trap formulation 2 open label, higher concentration
  Interventions: Biological: VEGF Trap

INTERVENTIONS:
Drug: VEGF Trap — VEGF Trap formulation 1, ITV-1
  Other Names: ITV-1
  Arms: ITV-1; ITV-2
Biological: VEGF Trap — VEGF Trap formulation 2 at higher concentration in Open label cohort
  Other Names: ITV-2
  Arms: ITV-2 OL

SUMMARY:
To assess the safety and tolerability of repeated intravitreal (ITV) administration of VEGF Trap.

DETAILED DESCRIPTION:
A double-masked study in which approximately 12 subjects will receive ITV injections of VEGF Trap every 4 weeks for a total of 3 doses. Once the subjects have received the 3 doses allowed in this study, they will be evaluated every 4 weeks for continued dosing of VEGF Trap for an additional 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Subfoveal CNV secondary to AMD.
* Central retinal (including lesion) thickness ≥ 250 µm as measured by OCT.
* ETDRS best-corrected visual acuity (BCVA) of 20/40 to 20/400 (73 to 20 letters)

Exclusion Criteria:

* No prior treatment with the following in the study eye:

  * Subfoveal thermal laser therapy;
  * Submacular surgery or other surgical intervention for the treatment of AMD;
  * Extrafoveal laser coagulation treatment within 12 weeks prior to Day 1 (Visit 2);
  * PDT or ITV administration of triamcinolone acetonide or any other steroid within 12 weeks prior to Day 1 (Visit 2);
  * Pegaptanib sodium within 8 weeks of Day 1 (Visit 2);
  * Juxtascleral steroids or anecortave acetate within 180 Days (6 months) prior to Day 1 (visit 2);
  * Prior systemic or intravitreal treatment with VEGF Trap or bevacizumab;
  * Any investigational agent for the treatment of eye disease within 12 weeks of Day 1 (Visit 2)
* History of any vitreous hemorrhage within 4 weeks prior to baseline injection visit.
* Aphakia or pseudophakia with the absence of a posterior capsule (unless it occurred as a result of a yttrium aluminum garnet [YAG] capsulotomy).
* Significant subfoveal atrophy or scarring.
* Any condition or laboratory abnormality that, in the opinion of the Investigator, would interfere with the assessment of disease status/progression or jeopardize the subject's appropriate participation in this study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10; Primary Completion 2007-09 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study will be safety and tolerability of the study treatment at Week 12 as assessed by ophthalmic examination and reporting of AEs. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Avner Ingerman, MD, Study Director — Regeneron Pharmaceutical
Locations (6):
- United States (6):
  - Fort Myers, Florida
  - Wichita, Kansas
  - Hagerstown, Maryland
  - Columbia, South Carolina
  - Austin, Texas
  - McAllen, Texas